CLINICAL TRIAL: NCT06056323
Title: A Phase I/II, Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of HB0045 in Patients With Advanced Solid Tumors
Brief Title: A Study of HB0045 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Gabrail Cancer Center Research (Other); Dana-Farber Cancer Institute (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0045-01; NCT05944276 (obsolete NCT alias)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Catalytic Domain

STUDY DESIGN:
Intervention Model Description: Phase I: Dose escalation with a conventional 3+3 design, including 1.5、5、15、30 and 40mg/kg dose group Phase II：Dose expansion phase. During the dose escalation process, expansion cohorts will be conducted based on the preliminary RP2D. A Simon 2-stage design will be utilized with a stopping rule to allow for early termination of a particular cohort at the end of Stage 1 if patients have insufficient responses to HB0045.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB0045 (Experimental): HB0045 IV every 3 weeks (q3w)
  Interventions: Drug: HB0045 Drug Product

INTERVENTIONS:
Drug: HB0045 Drug Product — Patients will be assigned to dose regimens in the order of enrollment and receive their assigned fixed dose of HB0045 via intravenous infusion, Q3W.
  Other Names: fixed dose combination of two antibodies targeting two different epitopes (N-terminal and catalytic site) of CD73

SUMMARY:
This is a phase I/II, open-label, multicenter study . During the study, subjects will be evaluated for safety, toxicity, tolerability, PK/PD, immunogenicity, biomarkers, and antitumor activity of HB0045. The phase I study will enroll up to 54 subjects with advanced solid tumors who have progressed on or after standard of care therapy and for whom there is no further treatment available that in the judgement of the patient's physician would be beneficial. One cycle is defined as 21 days.

DETAILED DESCRIPTION:
During the phase I study, the safety and tolerability of HB0045 will be evaluated in patients with advanced solid tumors including understanding of the preliminary efficacy. During this phase of the study, DLTs, MTD and MTD range will be observed which will inform RP2D. Phase I:Approximately 54 patients will receive HB0045 as a monotherapy at escalating doses.One cycle is defined as 3 weeks (21 days).

In the phase II study, the safety and preliminary efficacy of HB0045 at the RP2D will be evaluated in cohorts of patients with pancreatic, colorectal, ovarian cancer and/or other solid tumors.Phase II:During the dose escalation process, expansion cohorts will be conducted based on the preliminary RP2D.A Simon 2-stage design will be utilized with a stopping rule to allow for early termination of a particular cohort at the end of Stage 1 if patients have insufficient responses to HB0045. During Stage 1, 9 evaluable patients will be enrolled in each cohort; if no responses are observed within the cohort, then the cohort will be discontinued. If at least 1 response is observed, 8 additional evaluable patients will be enrolled in the cohort (Stage 2), for a maximum of 17 evaluable patients per cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years.
2. The subject can understand and willing to sign the ICF and is willing and able to comply with all study procedures.
3. Phase I: Patients with histologically or cytologically confirmed locally advanced, recurrent, or metastatic solid tumors (or clinically diagnosed hepatocellular carcinoma) that failed (progressed on or are intolerant of) all standard therapies known to provide clinical benefit; [These solid tumors include but not limited to: pancreatic, colorectal, ovarian, breast, lung, head and neck, prostate, renal cancer, and sarcoma, etc.]
4. Phase II: Patients who have had at least one systemic therapy and has progressed, and might benefit from the study drug in the Investigator's judgment, and have the following histological types (The types of tumors and the number of treatment lines may be adjusted based on phase I results and /or SRC discussions):

   a) Pancreatic cancer cohort: i. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma. ii. Unresectable, locally advanced recurrent or metastatic. b) CRC cohort: i. Histologically or cytologically confirmed colorectal cancer. ii. Molecular typing: non-dMMR/ non-MSI-H colorectal cancer. c) Ovarian cancer cohort: i. Histologically or cytologically confirmed unresectable metastatic ovarian, fallopian tube or peritoneal cancer ii. Epithelial type including high-grade serous cell carcinoma, endometrioid carcinoma or clear cell carcinoma.

   iii. No history of ileus (including signs or symptoms of ileus) within 3 months prior to screening.

   iv. Patients who had not received enterostomy within 3 months prior to screening.

   v. Have failed (progressed on or are intolerant of) all standard therapies known to provide clinical benefit; including but not limited to treatment with platinum-based chemotherapy if platinum-sensitive disease, and treatment with chemotherapy + bevacizumab if platinum-resistant and have not received prior bevacizumab.

   d) Other advanced cancer cohort(s): Tumor specific type that demonstrated partial response to HB0045 in dose escalation phase.
5. At least one measurable lesion as per RECIST v. 1.1 defined as non-nodal lesions having at least one dimension with a minimum size of 10 mm in the longest diameter by CT or MRI scan or ≥15 mm in short axis for nodal lesions. Radiographic disease assessment at baseline can be performed up to 21 days prior to the first dose.

   Note: Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
7. Life expectancy ≥12 weeks.
8. Patients with active hepatitis B virus (HBV) without active disease (HBV DNA titer <1000 cps/mL or 200 IU/mL), or who are cured of hepatitis C virus (HCV) with a negative HCV RNA test may be enrolled at the investigator's discretion.
9. Patients with known human immunodeficiency virus (HIV) infection and a cluster of differentiation 4 (CD4) count that is documented to be ≥350 cells/mm3 within 12 months before study screening, and if HIV-infected patients with a lower CD4+ count (<350cell/ mm3)，should be eligible only if they have a potentially curable malignancy or for interventions in a later stage of development that have demonstrated prior activity with a given cancer.
10. Adequate organ function within 14 days of the first dose as defined by the following criteria:

    1. Hematology i. absolute neutrophil count (ANC) ≥ 1.5×109/L ii. platelets (PLT) ≥ 100×109/L iii. hemoglobin (HGB) ≥ 90 g/L Note: The above items require that patients have not received any blood component or supportive therapy with growth hormones within two weeks prior to blood sampling.
    2. Renal function: Calculated creatinine clearance (CrCL) > 30 mL/min (Cockroft-Gault Equation)
    3. Liver function i. AST and ALT ≤ 2.5×ULN; AST or ALT ≤ 5×ULN if liver metastases are present ii. Total bilirubin (TBIL) ≤ 1.5×ULN; ≤3 X ULN for patients with Gilbert's disease
    4. Coagulation function i. International normalized ratio (INR) or prothrombin time (PT)≤ 1.5×ULN (unless the patient is on stable dose of oral anticoagulant) ii. Activated partial thromboplastin time (APTT)≤ 1.5×ULN
11. Women of childbearing potential must confirm a negative serum pregnancy test within 3 days prior to the initiation of study treatment and begin use of an effective birth control directly after testing negative for pregnancy; Fertile patients and their partners must agree to use acceptable contraception for the duration of study drug use and for 120 days after the last administration of study treatment.

    Acceptable contraception Single method i. Intrauterine device (IUD) ii. Vasectomy of a female subject's male partner iii. Contraceptive rod implanted into the skin Combined method (requires the use of two of the following) i. Diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide) ii. Cervical cap with spermicide (nulliparous women only) iii. Contraceptive sponge (nulliparous women only) iv. Male condom or female condom (cannot be used together) v. Hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin -only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection.
12. Recovery to Grade 0-1 from adverse events (AEs) related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, and endocrinopathies controlled with hormone replacement therapy.

Exclusion Criteria:

1. Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma. Patients with prostate cancer that is under active surveillance are eligible.
2. Have clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain or meningeal metastases may participate and be eligible for treatment provided they are stable and asymptomatic. Patients with asymptomatic brain or meningeal metastasis or patients who are symptomatically stable after treatment and are on≤ 10 mg/d prednisone or equivalent are eligible.
3. Cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure occurred within 6 months before study admission; QT-interval corrected according to Fridericia's formula (QTcB) > 480 milliseconds (ms) obtained from three consecutive ECGs; uncontrolled arrhythmia < 3 months of study entry (judged by the Investigator). Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.
4. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
5. Patients who have previously received allogeneic stem cell or solid organ transplantation.
6. History of severe allergic reactions, grade 3-4 allergic reactions to treatment with another monoclonal antibody or known to be allergic to protein drugs or recombinant proteins or excipients in HB0045 drug formulation.
7. History of Grade 3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for Grade 3 endocrinopathy that is managed with hormone replacement therapy).
8. Use of systemic corticosteroids in a dose equivalent to ≥10 mg/day of prednisone or other immunosuppressive agents < 2 weeks prior to screening; the use of topical, intraocular, intraarticular, intranasal, or inhaled corticosteroids and systemic steroids to prevent (e.g., allergy to contrast agents) or treat non-autoimmune condition (e.g., delayed hypersensitivity caused by exposure to allergens), or short course (< 5 days) will be allowed.
9. Have received antibiotics lasting over 1 week within 28 days prior to first dose.
10. Have received or will receive a live vaccine within 4 weeks prior to the first dose.
11. Any of the following infections

    1. Positive COVID-19 qRT-PCR or rapid screening test during screening; can be eligible after quarantine (14 days) if COVID-19 test becomes negative.
    2. Patients with active tuberculosis (TB) who are receiving anti-TB treatment or who received anti-TB treatment within 1 year prior to screening.
12. Prior treatment with agents targeting CD73 or A2AR.
13. Anticancer therapy < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (RT).
14. Major surgery (except for diagnostic needle biopsy or puncture and drainage or intravenous catheterization) or chemotherapy/ interventional therapy/radiation therapy/ablation therapy < 4 weeks prior to the first dose
15. Patients who have participated in any clinical trial of a drug or medical device within 4 weeks prior to the first dose.
16. Patients whose existing significant clinical abnormalities or laboratory abnormalities may affect the evaluation of the study drug by the Investigator's judgement. Psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up and affect patient's compliance or place the patient at high risk from treatment.
17. Other conditions which would make it inappropriate for the patient to participate as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Phase I: The incidence of Dose-Limiting Toxicities (DLTs) in patients receiving HB0045 | Up to 21 Days
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (3 weeks) of treatment.A Bayesian Logistic Regression Model (BLRM) based approach will be used to identify the set of HB0045 doses where the incidence of DLTs is no larger than 33%.
Phase I: Maximum Tolerated Dose(MTD) | Up to 36 Moths
  Maximum Tolerated Dose is defined as the highest dose in which the number of cases of DLT is less than 1/3 of the total patients in the first treatment cycle (DLT evaluation period) of the dose escalation phase.
  During the dose escalation phase of the study, if ≥33% DLTs occurred at a certain dose level, the maximum tolerated dose would be the dose level below that level, and if no ≥33% DLTs occurred after escalation to the highest dose, the highest dose will be considered MTD.
Phase II: Objective response rate (ORR) | Up to 24 Months
  ORR defined as the number of patients were confirmed complete response(CR) and/or partial response(PR) according to RECIST 1.1 divided by the patients with at least one tumour evaluation

SECONDARY OUTCOMES:
Anti-drug antibodies (ADA) | Up to 24 Moths
  Incidence of positive anti-drug antibodies(ADA).
Phase I＆II：Maximum serum concentration(Cmax) | within 48 hours after single HB0045 administered
  * Cmax refers to The maximum blood concentration of HB0045 after administration.
  * Sample concentration analysis method adopts ELISA .
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Phase I＆II：Half-life (t1/2) | within 3 months after first dose of HB0045 administered
  * t1/2 refers to the time of a half reduction of total drug concentration in the body.
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Phase I＆II：time of maximum concentration(Tmax) | within 3 months after first dose of HB0045 administered
  * Cmax, ss refers to The maximum blood concentration of HB0045 after four cycles administration.
  * Sample concentration analysis method adopts ELISA .
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Phase I＆II：Maximum serum concentration(Cmax,ss) | within 3 months after first dose of HB0045 administered
  * Cmax, ss refers to The maximum blood concentration of HB0045 after four cycles administration.
  * Sample concentration analysis method adopts ELISA .
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Phase I＆II：Half-life (t1/2, ss) | within 3 months after first dose of HB0045 administered
  * t1/2, ss refers to the time of a half reduction of total drug concentration in the body after four cycles of administration of HB0045.
  * parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Phase I＆II：time of maximum concentration(Tmax, ss) | within 3 months after first dose of HB0045 administered
  Peak time after HB0045 administration. The parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis
Phase I＆II：Area under the curve (AUC0-t） | Up to 24 Months
  AUC0-t refers to Area under the curve (AUC) from zero up to definite time t with extrapolation of the terminal phase.
  Parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis.
Phase I＆II：Area under the curve (AUC0-∞） | Up to 24 Months
  Area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase.
  Parameters will be calculated by Phoenix WinNonlin version 8.3 using noncompartmental analysis.
Disease control rate (DCR) | Up to 24 Months
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 divided by the patients with at least one tumour evaluation
Duration of response (DOR) | Up to approximately 2 years
  DOR defined as time from the first record of CR or PR to the first record of disease. DOR as evaluated by investigators according to RECIST v1.1.
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first)
Up to approximately 2 years | up to 2 years
  Overall survival is defined as the time from the start of treatment with HB0045 until death due to any cause. OS as evaluated by investigators according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yongmin Yang, Study Chair — Shanghai Huaota Biopharmaceutical Co., Ltd.
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Gabrail Pharmacology Phase 1 Research Center LLC, Canton, Ohio
  - UT M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No